CLINICAL TRIAL: NCT03193320
Title: Intraoperative Fluid Therapy Management in Low-risk Patients Under General Anesthesia- a Randomized Controlled Trial Comparing Liberal, Restrictive and Pleth Variability Index (PVI)-Guided Fluid Administration in a Day Surgery Setting
Brief Title: Management of Intraoperative Fluids in Ambulatory Surgery
Acronym: MIFAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Policlinica Metropolitana (Industry)
Responsible Party: Principal Investigator, Renzo Di Natale, Medical doctor (MD), Policlinica Metropolitana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1701
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia, General; Fluid Therapy; Ambulatory Surgical Procedures
Keywords: plethysmographic variability index; PVI

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be under general anesthesia during the interventions. Outcome assessors (nurses) will be blinded to the treatment provided in the operating rooms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liberal group protocol (Active Comparator): Fluid loading with 500 ml at induction. Baseline fluid infusion - 8 ml/kg/h. Fluid challenge - if mean arterial pressure (MAP) falls to < 65 mmHg, a fluid challenge will be administered.
  Interventions: Other: Fluid therapy protocol
- Restrictive group protocol (Active Comparator): No fluid loading at induction. Baseline fluid infusion - 4 ml/kg/h. Fluid challenges - if mean arterial pressure (MAP) falls to < 65 mmHg, a fluid challenge will be administered.
  Interventions: Other: Fluid therapy protocol
- PVI-guided group protocol (Experimental): No fluid loading at induction. Baseline fluid infusion - 2 ml/kg/h. PVI will be monitored continuously since anesthesia induction. Fluid challenges - if PVI rises >=13 (or MAP falls < 65 mmHg), a fluid challenge will be administered.
  Interventions: Other: Fluid therapy protocol

INTERVENTIONS:
Other: Fluid therapy protocol — Only ringer lactate (RL solution will be used). 1. Fluid loading at induction with 500 ml of ringer lactate solution will be given to some groups. 2. Base infusion rate varies according to group. 3. Fluid challenges - infusion of 250 ml over 5 min, a hemodynamic parameter specific to each group will be monitored for 10 min after the end of infusion to look for changes. Patients who do not respond to four (4) fluid challenges (volume infused 1000 ml) will be excluded.

SUMMARY:
This is a single-center prospective randomized control trial (RCT) to determine whether the continuous monitoring of the plethysmographic variability index (PVI) during low-risk surgeries, can be used to optimize the intraoperative fluid administration. Low-risk patients that attend our day surgery unit, and who will be operated under general anesthesia, will be randomized to either a liberal fluid group, a restrictive fluid group or a dynamic monitoring group (PVI-directed). The amount of fluid infused together with the time to discharge, will be assessed in each participant during the postoperative period along with additional secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* participants attending the unit for a day surgery procedure
* participants whose surgeries will be performed under general anesthesia
* aged between 18-65 years
* no abnormal findings on chest x-ray or electrocardiogram on preoperative evaluation
* patients undergoing procedures which do not require opening of the abdominal or thoracic cavities

Exclusion Criteria:

* ASA score III or higher
* patients undergoing surgeries which require additional pain management procedures (e.g. selective nerve blockade, epidural anesthesia, etc.)
* known pregnant women
* known kidney disease (or serum creatinine >1.8 mg/dl)
* known liver disease (or AST/ALT >60 U/l)
* known chronic heart failure (determined by a LVEF <55%)
* participants who develop hypotension intraoperatively and do not respond to 4 fluid challenges (1000 ml), requiring aggressive fluid resuscitation OR vasopressors
* estimated blood loss during surgery >250 ml
* development of an adverse reaction to any of the drugs administered during surgery (requiring additional medical management)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Total volume of fluid infused intraoperatively | 0 min after extubation
  Total volume of ringer lactate solution infused intraoperatively to participants (ml).
Time to discharge | 240 min after extubation (discharge)
  Time in hours (h) from anesthesia reversal to fulfillment of patient discharge criteria. Patients will be assessed by an attending nurse every 30 min to assess the fulfillment of these criteria.

SECONDARY OUTCOMES:
Significant postoperative nausea and vomiting (PONV) | 240 min after extubation (discharge)
  Presence of significant PONV as determined by a score ≥5 on the scale proposed by Myles SA et al. (BJA 2012)
Postoperative dizziness | 30 min after reversal
  Presence of patient self-reported dizziness in the post-operative period.
Postoperative fatigue | 30 min after reversal
  Presence of patient self-reported fatigue after surgery.
Postoperative thirst | 30 min after reversal
  Presence of patient self-reported thirst after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pascual M Carucci, MD, Study Director — Policlinica Metropolitana
Locations (1):
- Policlinica Metropolitana, Caracas, Miranda, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided